CLINICAL TRIAL: NCT05563597
Title: Cognitive Monitoring in Planned Arthroplasty Surgery
Acronym: COMPASS
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: Torbay and South Devon NHS Foundation Trust (Other); Claremont Medical Practice, Exmouth (Unknown); Peninsula Collaboration for Leadership in Applied Research and Care (PenCLAHRC) (Unknown); Peninsula Public Involvement Group (PenPIG), a division of PenCLAHRC (Unknown); South West Anaesthesia Research Matrix (SWARM) (Unknown); The Rame Group Practice, Torpoint (Unknown); Wesnes Cognition Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17/P/166
Record Dates: First submitted 2019-07-09; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2019-07

CONDITIONS: Cognitive Change

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Feasibility study testing a prospective observational methodology to assess the feasibility of serial remote monitoring of cognition with CogTrack™, an online cognitive assessment tool.

DETAILED DESCRIPTION:
A feasibility study testing a prospective observational methodology at two secondary care sites (Derriford Hospital, University Hospitals Plymouth NHS Trust and Torbay Hospital, Torbay and South Devon NHS Foundation Trust) and open to interested primary care practices (who refer patients to secondary care).

Serial cognitive testing will be performed using CogTrack™, a validated online cognitive assessment tool, over approximately an 11-week period. CogTrack™ requires two practice sessions to familiarise participants13, so the baseline CogTrack™ score will be that which is performed on the third occasion. Surgical patients will be tested both pre- and post-operatively. Non-surgical patients will have the assessments done at times to mirror those in the surgical group.

Target is to recruit 150 participants in the surgery group and 50 control patients from primary care.

The demographics and other data will be directly entered onto a secure electronic eCRF by a member of the research team. Only networked trust computers will be used and data entered onto a password protected database held on a shared network drive.

ELIGIBILITY:
Inclusion Criteria:

* Secondary Care (cases)
* Age over 60 years
* Listed for elective hip replacement
* Listed for elective knee replacement
* Able to consent for surgery
* Primary Care (controls) matched population by age

Exclusion Criteria:

* Patient refusal
* Operation in the previous 12 months
* Patients lacking capacity to sign their own consent form for surgery
* Patients already with a diagnosis of dementia or deemed to lack capacity
* Operation date within 3 weeks

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 60 undergoing elective hip or knee joint replacement surgery plus volunteer controls from primary care.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of patients approached | 18 months
  Number of patients approached
Number of patients recruited | 18 months
  Number of patients recruited
Number of patients declining | 18 months
  Number of patients declining
Number of withdrawals plus reason if given | 18 months
  Number of withdrawals plus reason if given
Completion rate of remote cognitive assessment | 18 months
  Completion rate of remote cognitive assessment
Completion rate of secondary assessment | 18 months
  Completion rate of secondary assessments
IT accessibility | 18 months
  IT accessibility
Acceptability questionnaire | 18 months
  Acceptability questionnaire

SECONDARY OUTCOMES:
Cognitive assessment | 18 months
  CogTrack™ :
  * This is an online validated tool to assess cognition that takes approximately 20 minutes to deliver and can be done remotely by the patient provided they have a computer with keyboard that can connect to the internet.
  * The first two assessments done will be training for the patient to gain familiarity and will not count as study data.
  * Scores are returned in 9 relevant domains
  * Attention Intensity Index, a composite score of reaction times from 3 different tasks will be the primary quantitative endpoint
  * Scores are not released to the patient or the assessor: results are uploaded to a secure database under a unique study code. Therefore, data will remain anonymous to the researchers of Wesnes Cognition Ltd. However, the clinical research team will be able to link the data to demographic and other data collected. Password protection on all databases maintains confidentiality at all times.
3D-CAM scores: | 18 months
  * To detect patients with delirium
  * The confusion assessment method (CAM)1 is widely adopted as a validated way to diagnose delirium, including in the post-operative period. However, in the clinical setting it can be challenging to deliver due to requirement of interviewer training and variation in application.
  * A new 3-minute diagnostic assessment, the 3D-CAM, has been developed and validated as a diagnostic assessment with high sensitivity and specificity for delirium.
  * It is important to identify those patients with delirium as this is often short-lived but may have longer term consequences.
  Tools scale consists of delirium being present or absent
Short form of the Informant Questionnaire on Cognitive Decline in the Elderly (Short IQCODE)2: | 18 months
  * To detect patients with possible dementia
  * This is a widely used tool for the initial assessment of possible dementia. Each question on the IQCODE is scored from 1 to 5. A score of 3 means that the subject is rated on average as 'no change'. A score of 4 means an average of 'a bit worse'. A score of 5 an average of 'much worse'.
  The IQCODE result is achieved by adding the score for each question and dividing by the number of questions. For the short IQCODE, divide by 16.
  A cutting point of 3.31/3.38 for dementia achieves a balance of sensitivity and specificity.
Pain score: | 18 months
  * To categorise patients as potentially being distracted, or not, by pain from performing the CogTrack™ test
  * Pain may affect cognitive processes and motivation. Therefore, it is important to ascertain levels of pain that patients experienced during the study and how this has affected their activity.
  VAS score: 0 (no pain)- 10 (worst pain)
Opioid and sedative consumption in previous 6 hours: | 18 months
  * Opioids and sedatives may affect cognition and hence we will be collecting this information alongside the cognitive testing. Opioid consumption will be converted to oral morphine equivalent doses (Appendix 7). Analgesics tend to have their highest pharmacological activity for the first few hours after a dose, hence the 6 hour window
  * This information will be gathered as part of the online CogTrack™ assessment using a free text box for participants to enter the drugs and doses they have taken in the preceding 6 hours
  * It is important this information is collected at each CogTrack™ assessment
Mood: | 18 months
  * Mood may affect someone's motivation and ability to do some of the assessments
  * We will therefore include a simple validated scale of mood, which will form part of the CogTrack™ cognitive assessment.
  * This is quick to complete and by having it as part of the online package it reduces burden on patients as well as researchers.
Single question of subjective memory deterioration: | 18 months
  o Assess how patients subjectively perceive any cognitive changes when compared to objective measures.
Clock drawing test (semi quantitative, score out of 3): | 18 months
  o Clock drawing has been used extensively in the study of cognitive changes. It assesses a range of cognitive functions, is relatively quick to administer (approximately 5 minutes) and acceptable to patients.
  A score of 0-3 is given depending of the presence of certain features of the performed task.
  Scale of marking 0-3

CONTACTS AND LOCATIONS:
Overall Officials: Gary Minto, Study Chair — University Hospital Plymouth NHS Trust
Locations (1):
- Torbay and South Devon NHS Trust, Torquay, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers